CLINICAL TRIAL: NCT03533270
Title: Urological Outcome of Posterior Urethroplasty in Patients With Pelvic Fracture and Urethral Distraction Defect in Assuit University
Brief Title: Urological Outcome of Posterior Urethroplasty in Patients in Assuit University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelkader, Dr., Assiut University
Other Study IDs: uretheroplasty
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Trauma;Pelvis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urethroplasty: Patients with traumatic urethral injury associated with pelvic fractures who underwent urethroplasty
  Interventions: Procedure: Urethroplasty

INTERVENTIONS:
Procedure: Urethroplasty — Surgical repair of Urethral injury

SUMMARY:
The management of posterior urethral disruption secondary to blunt pelvic injury remains controversial. While many groups have recommended early realignment of urethral distraction injuries, Classic reports advocate a suprapubic cystostomy at the time of injury with delayed, perineal approach urethral re- construction 4 to 6 months after injury . Timing of the intervention typically is classified as :

1. -Immediate treatment: when it takes place less than 48 hours after injury,
2. -Delayed primary treatment : after 2 to 14 days, and
3. -Deferred treatment : 3 months or more after injury.

DETAILED DESCRIPTION:
It is important to make a distinction between posterior urethral stricture and a pelvic fracture urethral distraction defect. Urethral stricture indicate a narrowing of the urethral continuity due to either instrumentation or partial urethral tears. In urethral distraction defects there is a gap between the membranous urethra and the bulbar urethral end. A distraction injury also involve all or any portion of the membranous urethra.

The management of posterior urethral disruption secondary to blunt pelvic injury remains controversial. While many groups have recommended early realignment of urethral distraction injuries, Classic reports advocate a suprapubic cystostomy at the time of injury with delayed, perineal approach urethral re- construction 4 to 6 months after injury. Timing of the intervention typically is classified as :

1. -Immediate treatment: when it takes place less than 48 hours after injury,
2. -Delayed primary treatment : after 2 to 14 days, and
3. -Deferred treatment : 3 months or more after injury.

Immediate open repair of posterior urethral injuries is usually associated with a higher incidence of strictures, re-stenosis, incontinence and impotence. Difficulty in identifying structures and planes as a result of hematoma formation and edema also hamper adequate mobilization and subsequent surgical apposition.

Contemporary urethral realignment employs actual realignment by fluoroscopic and endoscopic guidance of flexible cystoscopes that keep the urethral ends in the same cephalocaudad axis, followed by Seldinger technique catheter placement. The urethral catheter, which is usually maintained for 4 to 6 weeks, acts as a guide that allows the distracted urethral ends to come together as the pelvic hematoma slowly resorbs.

In the unstable or multisystem trauma patient, realignment often is delayed a few days to weeks (typically 2 to 14 days). the patient is managed by damage control and resuscitated in the intensive care unit while the urine is diverted by suprapubic tube placement first. Once the patient is stable, delayed urethral realignment is performed. Endourologic and radiologic techniques for realignment, theoretically, should not affect potency or urinary continence because no manipulation occurs of the periprostatic tissues or neurovascular bundles.

Types of surgical repair employed in posterior urethral distraction defect are 1) anastomotic urethroplasty, 2) Buccal mucosal urethroplasty, 3)Scrotal or penile island and 4) Johansen's urethroplasty. We aim to compare the outcomes of different management approachs for patients with posterior urethral distraction injuries after pelvic fractures in Assiut University Hospitals.

Aim of the work To evaluate outcomes of posterior urethroplasty in patients with pelvic fractures and posterior urethral distraction defect according to different patient characteristics (Age, prior manipulation), type of injury (type of fracture, gap length) and time of intervention.

ELIGIBILITY:
The inclusion criteria are:

All patients with pelvic fracture and urethral distraction injury (PFUDDI) except patients with any of the exclusion criteria.

The exclusion criteria are:

1. Bladder neck injury
2. Rectal injury
3. Urethrorectal injury
4. Spinal cord injury
5. Associated anterior urethral strictures

Min Age: 1 Year | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — No, Gender eligibility is based on biological gender identity
Study Population: Male patients underwent surgical repair of post traumatic urethral injury
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Presence of lower urinary tract symptoms | 1 year
  eg, hesitancy, frequency, obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Medhat El Hawary, MD, PhD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No